CLINICAL TRIAL: NCT02356289
Title: Safety, Tolerability, Preliminary Pharmacokinetics and Pharmacodynamics of Single Ascending Oral Doses of MYK-461 in Healthy Volunteers
Brief Title: Single Ascending Dose Study of MYK-461 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MyoKardia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MYK-461-002
Record Dates: First submitted 2015-02-02; First posted 2015-02-05 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — MYK-461

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MYK-461 (Experimental): single-dose, tablet formulation
  Interventions: Drug: MYK-461
- Placebo (Placebo Comparator): single-dose, tablet formulation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: MYK-461
  Arms: MYK-461

SUMMARY:
The purpose of this study is to establish initial safety, tolerability, pharmacokinetics and pharmacodynamics of MYK-461 in human subjects. This is a randomized, double-blind, placebo-controlled, sequential group, single ascending (oral) dose study in healthy volunteers aged 18-55 years.

ELIGIBILITY:
Inclusion Criteria:

* Normal body mass index (BMI)
* Normal LVEF
* Normal electrocardiogram (ECG)
* Females must not be breastfeeding and must be permanently sterilized or are postmenopausal.

Exclusion Criteria:

* Any structural abnormalities on echocardiography
* Positive results of HIV test and/or seropositive for HCV or HBV.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | 28 Days

SECONDARY OUTCOMES:
Determination of pharmacokinetics parameters | 28 Days
  maximum concentration (Cmax)
Determination of pharmacokinetics parameters | 28 Days
  time of the maximum measured concentration (Tmax)
Determination of pharmacokinetics parameters | 28 Days
  area under the concentrationtime curve (AUC)
Determination of pharmacokinetics parameters | 28 Days
  half-life (t1/2)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan C Fox, MD, PhD, Study Director — MyoKardia, Inc.
Locations (1):
- Quintles LTD, London, United Kingdom